CLINICAL TRIAL: NCT03683862
Title: Objective Evaluation of Compliance After Orthodontic Treatment Using Thermoplastic or Hawley Retainers: A Randomized Controlled Trial
Brief Title: Compliance After Orthodontic Treatment Using Thermoplastic or Hawley Retainers
Acronym: OrthoComply
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Despina Koletsi, Researcher, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 341/10.07.17
Record Dates: First submitted 2018-09-23; First posted 2018-09-25 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Orthodontic Retention Compliance
Keywords: hawley; thermoplastic; orthodontic retention; compliance; vacuum- formed
MeSH Terms: conditions — Patient Compliance | interventions — Orthodontic Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoplastic Retainer (Experimental): Impressions of the upper arch will be taken at the day of bracket debonding and the retainer will be delivered in 24 hours. TheraMon microchip will be embedded within the appliance and patients will be instructed to wear the appliance 24 hours/ day.
  Interventions: Other: orthodontic appliance
- Hawley Retainer (Active Comparator): Impressions of the upper arch will be taken at the day of bracket debonding and the retainer will be delivered in 24 hours. TheraMon microchip will be embedded within the appliance and patients will be instructed to wear the appliance 24 hours/ day.
  Interventions: Other: orthodontic appliance

INTERVENTIONS:
Other: orthodontic appliance — Orthodontic device for retention in the upper arch, after the end of orthodontic treatment

SUMMARY:
This study aims to assess adolescent's compliance after the end of orthodontic treatment using either thermoplastic or Hawley retainers in the upper arch, with the aid of TheraMon microsensor (MC Technology GmbH).

ELIGIBILITY:
Inclusion Criteria:

* patients that have completed orthodontic treatment (are at stage of debonding) with fixed appliances in the upper and lower arch
* age 12- 18

Exclusion Criteria:

* systematic diseases
* craniofacial anomalies (clefts, etc)
* handicapped patients with problems of compliance
* pregnant women
* previous orthodontic treatment or compromise orthodontic treatment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Compliance of retainer wear | 3 months
  Compliance of retainer wear at 3 months, as expressed by average hours of daily wear (with the aid of TheraMon)

SECONDARY OUTCOMES:
Compliance of retainer wear | 1 month
  Compliance of retainer wear at 1 month, as expressed by average hours of daily wear (with the aid of TheraMon)
Association between objective compliance assessment and diary reported hours | 3 months
  Association between objective compliance assessment (TheraMon) and diary reported hours (by patient)
Association between objective compliance assessment and diary reported hours | 1 month
  Association between objective compliance assessment (TheraMon) and diary reported hours (by patient)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Vagdouti, Principal Investigator — School of Dentistry, National and Kapodistrian University of Athens
Locations (1):
- School of Dentistry, Department of Orthodontics, National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vagdouti G, Karvouni E, Bitsanis E, Koletsi D. Objective evaluation of compliance after orthodontic treatment using Hawley or vacuum-formed retainers: A 2-center randomized controlled trial over a 3-month period. Am J Orthod Dentofacial Orthop. 2019 Dec;156(6):717-726.e2. doi: 10.1016/j.ajodo.2019.07.008. PMID 31784005